CLINICAL TRIAL: NCT03335774
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group Study to Evaluate Safety and Efficacy of 25 mg Hydrocortisone Acetate Suppositories in the Treatment of Symptomatic Internal Hemorrhoids.
Brief Title: Evaluate Safety and Efficacy of 25 mg Hydrocortisone Acetate Suppositories in Treatment of Internal Hemorrhoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nivagen Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDCS 1701 (formerly 1-2017)
Record Dates: First submitted 2017-10-30; First posted 2017-11-08 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Internal Hemorrhoids
MeSH Terms: interventions — Suppositories

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone Acetate Suppository, 25 mg (Active Comparator): One (1) Hydrocortisone Acetate Suppository, 25 mg is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
  Interventions: Drug: Hydrocortisone Acetate Suppository, 25 mg (Nivagen)
- Placebo (Vehicle) Suppository (Placebo Comparator): One (1) Placebo (Vehicle) Suppository is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
  Interventions: Drug: Placebo (Vehicle) Suppository (Nivagen)

INTERVENTIONS:
Drug: Hydrocortisone Acetate Suppository, 25 mg (Nivagen) — One (1) Hydrocortisone Acetate Suppository, 25 mg is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
  Arms: Hydrocortisone Acetate Suppository, 25 mg
Drug: Placebo (Vehicle) Suppository (Nivagen) — One (1) Placebo (Vehicle) Suppository is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
  Arms: Placebo (Vehicle) Suppository

SUMMARY:
A randomized, double-blind, placebo-controlled, multicenter, parallel group study of the safety and efficacy of Hydrocortisone Acetate Suppositories, 25 mg compared to placebo suppositories in the treatment of symptomatic internal hemorrhoids.

DETAILED DESCRIPTION:
STUDY DESIGN:

25 mg hydrocortisone suppositories administered twice daily compared to a vehicle placebo in approximately 100 subjects with symptomatic internal hemorrhoids. Subjects will be randomized in a 1:1 ratio (Test product: placebo).

The study will consist of 2 periods:

1. Treatment Period (2 weeks/ Days 1-14)
2. Follow-up Period (2 weeks/ Days 15-28)

The visits are as follows:

Visit 1 (Day 1 Baseline/Randomization) Visit 2 (Day 8±1, Interim Visit) Visit 3 (Day 15±2, End of Treatment Visit) Visit 4 (Day 29±3, End of Study Visit)

ENDPOINTS:

1. Clinician Reported Outcome (ClinRO) - Anoscopy (Visits 1, 3). Anoscopy - Visual assessment of hemorrhoids. Video of the procedure will be recorded for blinded central reading and assessment
2. Patient Reported Outcome: Subjects will use Daily Diaries to record the time and date of each medication application, concomitant medication and adverse events. The subjects will complete the Subject Questionnaire at Visits 1, 2, 3 and 4 (or early termination) and daily between visits.

ELIGIBILITY:
Inclusion Criteria:

* internal hemorrhoids.
* hemorrhoidal bleeding.
* male or female aged 18 years and older.
* willing to forego the use of non-prescription (OTC) and prescription medication or procedures for the treatment of hemorrhoidal disease and/or pain for the duration of the study.
* agree to not change their diet during the study.

Exclusion Criteria:

* external hemorrhoids.
* using other OTC or prescription medications for treatment of hemorrhoidal disease and/or pain.
* pregnant or nursing female.
* received systemic glucocorticoids within the last 2 months prior to starting study.
* participated in an investigational drug study within 30 days prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Shukla, MS, MBA,, Study Director — Nivagen Pharmaceuticals
Locations (2):
- Clinical Research, Charlotte, North Carolina, United States
- Clinical Research, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nivagen Pharmaceuticals Inc. — http://www.nivagen.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mostly patients were recruited from the existing database
Groups:
- Hydrocortisone Acetate Suppository, 25 mg: One (1) Hydrocortisone Acetate Suppository, 25 mg is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
  Hydrocortisone Acetate Suppository, 25 mg: One (1) Hydrocortisone Acetate Suppository, 25 mg is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
- Placebo (Vehicle) Suppository: One (1) Placebo (Vehicle) Suppository is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
  Placebo (Vehicle) Suppository: One (1) Placebo (Vehicle) Suppository is inserted into the anal canal twice daily (morning and evening) for 2 weeks (14 days).
Period: Overall Study
Arm/Group | Hydrocortisone Acetate Suppository, 25 mg | Placebo (Vehicle) Suppository
Started | 51 | 52
Completed | 50 | 51
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone Acetate Suppository, 25 mg | Placebo (Vehicle) Suppository | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (15.43) | 50.8 (15.57) | 50.6 (15.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 31 | 27 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 22 | 46
  Not Hispanic or Latino | 27 | 30 | 57
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
  India | 21 | 22 | 43
Swelling of hemorrhoid [Mean (Standard Deviation); unit: scores on a scale] — At Baseline, objective measurement of swelling of hemorrhoids was conducted utilizing Anoscopy. Recorded Video was sent for blinded central reading and assessment, and rated as: No swelling, score of 0; Mild swelling : score of 1; Moderate swelling: score of 2; Severe swelling: score of 3; Very Severe swelling: score of 4
  scores on a scale | 2.9 (0.68) | 2.8 (0.60) | 2.85 (0.64)
Itching severity [Mean (Standard Deviation); unit: Scores on a scale] — During the baseline period, patient-reported outcome (PRO) associated with symptom of 'itching' was collated by deploying the Internal Hemorrhoid Sign and Symptom Assessment (IHSSA) questionnaire.
  The mean score from the Screening period was considered the baseline score. Itching was scored from on 0-4 scale (0 = No itching, 1 = A little itching, 2 = Moderate itching, 3 = A lot of itching, 4 = Worst itching) Population: 1 subject in each of treatment arms did not meet threshold compliance % of completing the PRO questionnaire, and hence could not be included in the analysis.
  Scores on a scale
    number analyzed (Participants) | 50 | 51 | 101
    (all) | 2.15 (0.49) | 2.12 (0.50) | 2.13 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Swelling
Description: Reduction in the swelling of internal hemorrhoid was measured by anoscopy. Visual assessment of hemorrhoids was performed at end of treatment. Video of the procedure will be recorded for blinded central reading and assessment. Swelling was graded on a scale from "0 - None" to "4 - Very Severe".
  Numeric grades and their changes from baseline are summarized descriptively by visit and treatment group. Changes from baseline will be compared between the treatment groups. Mean difference between the groups and its 95% confidence interval will be displayed at Visit 4, along with the p-value from the two-sample t-test.
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone Acetate Suppository, 25 mg | Placebo (Vehicle) Suppository
Number analyzed (Participants) | 50 | 51
scores on a scale | 2.3 (0.74) | 2.0 (0.68)
Statistical Analysis 1: Comparison: Hydrocortisone Acetate Suppository, 25 mg vs Placebo (Vehicle) Suppository; The statistical analyses were conducted using SAS software Version 9.4.All statistical tests were two-sided at a significance level of α = 0.05. Continuous data were presented using descriptive statistics (i.e. number of subjects, mean, SD, median, minimum, and maximum).Baseline value of each assessment was defined as the latest available assessment obtained prior to the first administration of the study drug; Test type: Superiority — To determine if the 'hydrocortisone' arm was indeed superior than 'placebo' to reduce swelling and itching associated with internal hemorrhoids; p = 0.8918, t-test, 2 sided

2. Primary Outcome: Reduction in Itching Severity
Description: Patient-reported outcome (PRO) was collated and analyzed by deploying the Internal Hemorrhoid Sign and Symptom Assessment (IHSSA) questionnaire. The patients updated the questionnaire on a daily basis between visits 1-5. Responses to each item were averaged across each period.
  The mean score from the Screening period was considered the baseline score.
  Mean scores and their changes from baseline were summarized.
  Itching was scored from on 0-4 scale (0 =No itching, 1 = A little itching, 2 =Moderate itching, 3 = A lot of itching, 4 = Worst itching that you could imagine
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone Acetate Suppository, 25 mg | Placebo (Vehicle) Suppository
Number analyzed (Participants) | 50 | 51
scores on a scale | 0.74 (0.56) | 0.71 (0.61)
Statistical Analysis 1: Comparison: Hydrocortisone Acetate Suppository, 25 mg vs Placebo (Vehicle) Suppository; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8323, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Total time period for which AE data was collected was ~6 weeks for each subject
Description: Hydrocortisone suppositories have been prescribed for 5 decades for the management of internal hemorrhoids. The formulation is expected to act locally, with negligible systemic absorption. Therefore, risk of SAEs and mortality are non-existent.
Arm/Group | Hydrocortisone Acetate Suppository, 25 mg | Placebo (Vehicle) Suppository
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 1/50 | 2/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone Acetate Suppository, 25 mg (N=50) | Placebo (Vehicle) Suppository (N=51)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Excess calclium

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03335774/Prot_SAP_001.pdf